CLINICAL TRIAL: NCT05839704
Title: Comparison of Bilateral Erector Spinae Plane Block Versus Serratus Anterior Plane Block Plus Subcostal Transversus Abdominus Plane Block for Bariatric Sleeve Gastrectomy Surgery: A Randomised Clinical Trial
Brief Title: A Comparison of Two Regional Techniques for Bariatric Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Dr David Cosgrave, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUIG-2023-001
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Bariatric Surgery Candidate; Weight Loss; Surgery
Keywords: Sleeve Gastrectomy; Regional Anaesthesia; Opioid Sparing Anaesthesia
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patient, care provider and primary investigator will not be blinded to the intervention. The outcomes assessor who collects the post operative data will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Erector Spinae Plane Block (Experimental): Patients in this arm will receive standard anaesthesia as per our bariatric anaesthesia protocol. They will also receive preoperative ultrasound guided bilateral single shot erector spinae plane blocks at the level of the 8th transverse process.
  Interventions: Procedure: Bilateral Erector Spinae Plane Block
- Abdominal Wall Blocks (Active Comparator): Patients in this arm will receive standard anaesthesia as per our bariatric anaesthesia protocol. They will also receive bilateral subcostal transversus abdominus plane blocks and a left sided serrratus plane block, postoperatively, while under general anaesthetic.
  Interventions: Procedure: Abdominal Wall Blocks

INTERVENTIONS:
Procedure: Bilateral Erector Spinae Plane Block — Patient will receive local ropivacaine 0.75% with lignocaine 1% with adrenaline, administered under ultrasound into the erector spinae plane at the level of T8.
  Arms: Bilateral Erector Spinae Plane Block
Procedure: Abdominal Wall Blocks — Patient will receive local ropivacaine 0.75% with lignocaine 1% with adrenaline, administered under ultrasound into the subcostal transversus abdominus plane bilaterally and the serratus plane on the left side
  Arms: Abdominal Wall Blocks

SUMMARY:
Regional anaesthetic techniques, or nerve blocks, are commonly used to provide postoperative pain relief for patients undergoing surgery. At present in University Hospital Galway, it is standard practice for patients undergoing bariatric sleeve gastrectomy surgery to receive a regional anaesthetic technique to improve their postoperative pain. There are a number of different regional anaesthetic options available for this surgery, but as yet, published evidence regarding which specific approach confers most benefit for patients is lacking. This study aims to compare two regional anaesthetic techniques - erector spinae plane blockade versus serratus anterior plane blockade plus subcostal transversus abdominus plane blockade - and assess if one approach provides a superior quality of recovery postoperatively for sleeve gastrectomy patients over the other.

DETAILED DESCRIPTION:
The World Health Organisation describes obesity as an excessive accumulation of fat that presents a risk to health. Obesity is commonly defined as a BMI of greater than 30.

Obesity is a growing public health concern worldwide, with WHO statistics estimated in 2016 that 650 million people worldwide were obese, and this figure is predicted to rise annually. Obesity is an independent risk factor for a myriad of medical conditions, including but not limited to type 2 diabetes mellitus, obstructive sleep apnoea, hypertension, hyperlipidaemia and ischaemic heart disease. Obesity is also a difficult condition to treat, involving lifestyle modifications, psychological therapies, medical management and surgery. Limited long-term success of behavioural and pharmacological therapies in serious obesity have led to increasing interest in bariatric surgery. Surgery is considered for those patients who are suffering from complications of obesity, are at high risk of morbidity and mortality and who have not achieved adequate weight loss with lifestyle modification and medical management. Bariatric surgery can result in very substantial weight loss, resolution of obesity-related comorbidities and greatly improved quality of life for patients. Successful treatment of obesity via bariatric surgery has been shown to eliminate type two diabetes mellitus in up to 80% of patients. Bariatric surgery has been similarly shown to improve or eliminate obstructive sleep apnoea, hypertension and gastroesophageal reflux disease.

During the past two decades, an increasing number of bariatric surgical procedures have been performed worldwide. The most prevalent procedures from 2000 - 2010 were gastric bypass or gastric banding surgeries. In the past decade however, laparoscopic sleeve gastrectomy has become increasingly popular. Sleeve gastrectomy is a permanent method of reducing the size of the stomach. The SLEEVEPASS (2018) and SM-BOSS (2018) trials conferred similar weight loss and improvement in comorbidities such as type 2 diabetes after sleeve gastrectomy when compared with gastric bypass, but with lower morbidity and mortality rates. Sleeve gastrectomy has also been shown to decrease concentrations of ghrelin, the human "hunger hormone", which may explain the reduction in hunger and rapid weight loss in many patients postoperatively. Unfortunately, bariatric surgery is frequently complicated by considerable postoperative pain, which can be difficult to manage. These patients often suffer from obstructive sleep apnoea and are at risk of respiratory dysfunction postoperatively, particularly when opioid analgesia is administered, with alternative analgesic methods preferred. The Guidelines for Perioperative Care in Bariatric Surgery, published in 2016, highlighted the successful use of regional analgesia techniques for bariatric surgical patients. The ERAS (Enhanced Recovery After Surgery) Society 2021 guidelines recommend opioid sparing analgesia, which is our current practice in UHG, with a note on lacking evidence regarding which specific regional anaesthesia approach is preferable. Several regional analgesic options exist, including serratus anterior plane block, transversus abdominis plane (TAP) block and quadratus laborum block. Abdominal wall blocks such as the transversus abdominus plane block have been investigated with equivocal results, likely in part because they provide only somatic analgesia. At present in University Hospital Galway, the method utilised for regional analgesia for the majority of laparoscopic sleeve gastrectomy surgery is a combination of both serratus anterior plane block and subcostal TAP block. The erector spinae plane block (ESB) is a relatively novel regional anaesthesia technique first described in 2016. A very limited number of studies to date have been performed regarding ESB in bariatric surgery, with early indications suggesting that it may provide an opportunity to provide increased postoperative analgesia in this cohort of patients. An extensive literature review revealed a total of four randomised trials investigating the efficacy of ESB in bariatric surgery patients. Two of these trials compare ESB vrs. no block, while two compare ESB vrs. TAP block. To date, there have been no clinical trials or case reports published comparing erector spinae plane block vrs the combination of both serratus anterior plane block and subcostal TAP block in laparoscopic sleeve gastrectomy patients. This study aims to contribute to filling this gap in the literature by examining quality of recovery postoperatively to establish whether there is a difference between analgesia provided by erector spinae plane block versus that provided by serratus anterior plane block + subcostal TAP block in this cohort of patients. Of note, all patients undergoing this surgery in UHG would usually receive a regional analgesia technique, regardless of their enrolment in this study. The aim of this study is to compare the two regional analgesia techniques to identify the more efficacious approach.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* Undergoing laparoscopic sleeve gastrectomy surgery
* Ability to provide written informed consent
* ASA grade I-III

Exclusion Criteria:

* Inability to provide informed consent
* Pre-existing infection at block site
* Severe coagulopathy
* Allergy to local anaesthesia
* Previous history of chronic pain condition
* Previous history of opioid dependence/abuse
* Predicted inability to cooperate with completion of QoR-15 score on postoperative day 1
* Postoperative admission to ICU for prolonged ventilation postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score at 24h | 24 hours after the block is administered
  The QoR-15 score will be taken by the outcome assessor on the post operative ward.

SECONDARY OUTCOMES:
Pain scores at rest and on movement | 24 hours after block administration
  Self reported pain scores using verbal rating scale
Time to first analgesia in recovery room | Immediate post op recovery up to 24 hours
  The time from end of surgery to first administration of analgesia in recovery
24hr opioid consumption | 24 hours post block administration
  Total opioid consumption in oral morphine equivalents will be recorded at 24 hours
Length of stay | 30 days
  The length of stay in hospital from surgery to ready to discharge
Incidence of PONV/use of antiemetic rescue; | 24 hours post block administration
  The self reported occurrence of any post operative nausea and vomiting and the total dose of antiemetics administered
Incidence and severity of postoperative complications using Comprehensive Complication Index calculator | 30 days post op
  The Comprehensive Complications Index Calculator will be used to assess for any complications related to surgery or anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Galway, Galway, Ireland

REFERENCES:
- [Derived] Wiseman PN, Van der Walt M, O'Riordan M, Brosnan K, Shaikh M, Cosgrave D. A comparison of efficacy of erector spinae plane block versus serratus anterior plane block plus subcostal transversus abdominus plane block for bariatric laparoscopic sleeve gastrectomy surgery: study protocol for a randomised clinical trial. Trials. 2024 Sep 28;25(1):634. doi: 10.1186/s13063-024-08472-4. PMID 39342346